CLINICAL TRIAL: NCT05301998
Title: Tridimensional Geometric Modeling of the Breast. Interest in Creating a Generic Biomechanical Model Useful for Simulation and Surgical Prediction
Brief Title: Tridimensional Geometric Modeling of the Breast
Acronym: SENO 3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL21_0525; 2021-A02539-32 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2022-02-25; First posted 2022-03-31 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Skin Elasticity
Keywords: 3D geometric model; Breast surgery; Breast MRI; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Other): Measurements of elasticity and thickness will be performed for each of the 200 patients.
  Among the 200 patients, 10 will have a breast MRI in 3 different positions
  Interventions: Other: Skin and thickness measurement/breast MRI

INTERVENTIONS:
Other: Skin and thickness measurement/breast MRI — Patient will be installed in dorsal decubitus position. Measurements will be performed at 3 sites on one breast: at the areola, above the areola and below. Measurements will be performed by a single gynecologist using a cutometer provided by TIMC-IMAG laboratory of Grenoble. Three measurements will be performed at each site. Duration of measurements will be approximately 15 minutes.
  Measurement of skin thickness will be performed using an ultrasound device available in obstetrics/gynecology consultation department. The measurement will be performed at 3 sites. The duration of the measurements will be of approximately 10 minutes.
  Among the 200 patients, 10 patients who should benefit from a breast MRI as part of their follow-up, will have a breast MRI in 3 different positions: prone (standard protocol) and two additional acquisitions (as part of the research) in dorsal and right lateral decubitus. This examination will be scheduled in the senology department of the Lapeyronie Hospital

SUMMARY:
The use of a personalized 3D model of the breast in the management of breast cancer would be very useful to help the surgeon better understand the three-dimensional location of tumors in the operative position and thus better plan incisions and dissection of the breast tissue. This could be achieved with the help of a 3D biomechanical breast model that ideally should integrate the patient-specific mechanical properties of all breast tissue structures. The elasticity of the skin and especially the consideration of factors that can make it vary with age has been little studied. However, the integration of this parameter would clearly increase the robustness of the 3D model.

Main objective:

To perform a pilot evaluation of the performance of the biomechanical model by integrating the biomechanical characteristics of the skin and the collagenous architecture of the breast, during the transition from prone to supine or lateral position.

Secondary Objectives:

To describe the values of skin elasticity and thickness at different points of the breast, in women in the general population To search for clinical factors predictive of elasticity and skin thickness To carry out a pilot description of the collagen architecture of the breast

Participation in this study will be offered to all patients consulting the gynecology-obstetrics department of the Montpellier University Hospital and meeting the inclusion criteria-Visit 1: Inclusion and measurement of skin thickness and elasticity:

Inclusion will take place during the follow-up consultation in the obstetrics gynecology department of the Montpellier University Hospital. The patient's written consent will be obtained after a reflection period at the end of the consultation. Measurements of elasticity and thickness will then be performed for each of the 200 patients. Skin elasticity: The patient will be installed in dorsal decubitus position, with her arms at her sides on an examination table. Measurements will be performed at 3 sites on one of the two breasts: at the areola, above the areola and below. The measurements will be performed by a single gynecologist in the gynecology department using a cutometer provided by a laboratory of Grenoble. It has just been used by the Dutch Cancer Institute in Amsterdam to measure the elasticity of the tongue in a clinical study including 10 patients. Three measurements will be performed at each site. One measurement corresponds to a 10-second suction time (progressive rise of the depression) followed by 5 seconds of relaxation of the measurement site.

The duration of these measurements will be approximately 15 minutes. Skin thickness: The measurement of skin thickness will be performed using an ultrasound device available in the obstetrics and gynecology consultation department. The measurement will be performed at 3 sites. The duration of the measurements will be of approximately 10 minutes. Adverse events will be collected at the end of the measurements.

-Visit 2: Within 3 weeks after the first visit. Among the 200 patients, 10 patients who should benefit from a breast MRI as part of their follow-up, will have a breast MRI in 3 different positions: prone (standard protocol) and two additional acquisitions (as part of the research) in dorsal and right lateral decubitus. This examination will be scheduled in the Lapeyronie Hospital.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in France. Its screening and diagnosis use mammography, ultrasound and MRI. These imaging only show the topography of the tumors in the breast volume in two dimensions (2D). The surgeon must then mentally reconstruct the three-dimensional (3D) anatomy of the breast before planning the surgery.The use of a personalized 3D model of the breast would be very useful to help the surgeon to better understand the three-dimensional localization of the tumors in the operative position and thus to better plan the incisions and the dissection of the breast tissue, preserving the maximum of healthy tissue but also being more relevant in the oncological aspect.

This could be achieved with the help of a 3D biomechanical model of the breast which should ideally integrate the subject-specific mechanical properties of all the tissue structures of the breast. However, obtaining a model of the breast is very difficult due to the complexity and diversity of the 3D geometry of the structures and their highly heterogeneous mechanical character. All breast tissues (skin, connective tissue, mammary gland, fat, pectoral muscle) must be modeled. For this, their mechanical behavior must be known. As biomechanical properties vary according to ex-vivo and in-vivo conditions, it is important to obtain in-vivo measurements.

The biomechanical properties of the breast skin have been little studied. The integration of the mechanical parameters of the skin would thus clearly increase the robustness of a 3D model.

Some studies have focused on skin elasticity, mainly on the arms and face. Several non-invasive measurement techniques of the biomechanical properties of the skin have been tested: suction test, torsion test, bi-axial test, and multi-axial test. These techniques may be dependent on the experimental conditions: tension application technique, probe size, skin thickness, ... Among these procedures, suction tests are considered as a reference technique, non-invasive and easy to use, for the measurement of skin elasticity.

The mobility and deformation of the breast skin make it difficult to obtain accurate measurements of biomechanical properties. Sutradhar et al studied these properties in 23 women: variations in elasticity were found for different regions of the breast; lying or standing did not appear to have an impact. In 2016, Coltman et al conducted a study on breast skin elasticity and thickness involving 339 women. Regarding factors that may influence skin elasticity, Coltman et al found a decrease in skin elasticity with age. This effect was not found in the study by Sutradhar et al. A study of 15 women showed a variation in skin elasticity of the breast according to the cycle and whether or not they were taking contraception.Main objective:

To perform a pilot evaluation of the performance of the biomechanical model by integrating the biomechanical characteristics of the skin and the collagenous architecture of the breast, during the transition from prone to supine or lateral position.

Secondary Objectives:

To describe the values of skin elasticity and thickness at different points of the breast, in women in the general population To search for clinical factors predictive of elasticity and skin thickness To carry out a pilot description of the collagen architecture of the breast

Participation in this study will be offered to all patients consulting the gynecology-obstetrics department of the Montpellier University Hospital and meeting the inclusion criteria-Visit 1: Inclusion and measurement of skin thickness and elasticity:

Inclusion will take place during the follow-up consultation in the obstetrics gynecology department of the Montpellier University Hospital. The patient's written consent will be obtained after a reflection period at the end of the consultation. Measurements of elasticity and thickness will then be performed for each of the 200 patients. Skin elasticity: The patient will be installed in dorsal decubitus position, with her arms at her sides on an examination table. Measurements will be performed at 3 sites on one of the two breasts: at the areola, above the areola and below. The measurements will be performed by a single gynecologist in the gynecology department using a cutometer provided by laboratory of Grenoble. It has just been used by the Dutch Cancer Institute in Amsterdam to measure the elasticity of the tongue in a clinical study including 10 patients. Three measurements will be performed at each site. One measurement corresponds to a 10-second suction time (progressive rise of the depression) followed by 5 seconds of relaxation of the measurement site.

The duration of these measurements (installation of the patient - installation of the material - realization of the measurements) will be approximately 15 minutes.

Skin thickness: The measurement of skin thickness will be performed using an ultrasound device available in the obstetrics and gynecology consultation department. The measurement will be performed at 3 sites. The duration of the measurements will be of approximately 10 minutes. Adverse events will be collected at the end of the measurements.

-Visit 2: Within 3 weeks after the first visit. Among the 200 patients, 10 patients who should benefit from a breast MRI as part of their follow-up, will have a breast MRI in 3 different positions: prone (standard protocol) and two additional acquisitions (as part of the research) in dorsal and right lateral decubitus. This examination will be scheduled in t the Lapeyronie Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Up to 18 years old
* Understanding and acceptance of the protocol

Exclusion Criteria:

* Person protected by law under guardianship or curatorship
* Failure to obtain free, informed and written consent after a reflection period
* A patient who is not a member or beneficiary of a national health insurance system
* Patient with a skin disease or a skin lesion
* Person deprived of liberty by judicial or administrative decision
* Application of a cream on the skin within 12 hours before the measurements

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Measurement of skin elasticity using a cutometer | At baseline
  Skin elasticity measurements will be taken at 3 sites on one of the two breasts, during their 1st visit (baseline): at the level of the areola, above the areola and below. They will be performed by a single gynecologist from the gynecology department. Measurements will be made using a cutometer. It includes a computer, tubing connected to a 10, 15 or 20 mm cup. Three measurements will be carried out on each of the sites. A measurement corresponds to a time of gradual rise in suction of 10 seconds followed by 5 seconds of relaxation of the measurement site.
  A method based on an inverse model will then make it possible to estimate the local elasticity (Young's modulus) of the skin.
Measurement of skin thickness using an ultrasound device | At baseline
  Measurements of skin thickness will be made using an ultrasound machine available in the gynecology department. They will be done at 6 sites on one of the two breasts, during their 1st visit (baseline).
Collagen architecture of the breast | 3 weeks after baseline
  Precise 3D anatomical description of different breast tissues, the position and orientation of the tissues, on 10 patients with additional MRI acquisitions, at the 2nd visit (3 weeks after the 1st visit).
3D model | Through study completion, an average of 1 year
  To carry out a pilot evaluation of the performance of the biomechanical model by integrating the biomechanical characteristics of the skin and the collagenous architecture of the breast, during the transition from the prone position to the dorsal or lateral decubitus position

SECONDARY OUTCOMES:
Age in years | At baseline
  Evaluate the potential predictive factors of the biomechanical characteristics of the skin.
Body Mass Index in kilogram per square meter | At baseline
  Evaluate the potential predictive factors of the biomechanical characteristics of the skin.
Bra cup size | At baseline
  Evaluate the potential predictive factors of the biomechanical characteristics of the skin.
Time in the menstrual cycle | At baseline
  Evaluate the potential predictive factors of the biomechanical characteristics of the skin.
Contraception | At baseline
  Presence and type of contraception. Evaluate the potential predictive factors of the biomechanical characteristics of the skin.
Menopausal status | At baseline
  Evaluate the potential predictive factors of the biomechanical characteristics of the skin.
History of breast radiotherapy | At baseline
  Evaluate the potential predictive factors of the biomechanical characteristics of the skin.
Breastfeeding history | At baseline
  Breastfeeding history after their potential pregnancies. Evaluate the potential predictive factors of the biomechanical characteristics of the skin.
History of breast surgery | At baseline
  Evaluate the potential predictive factors of the biomechanical characteristics of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Martha DURAES, MD, Study Director — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, Outside of the US, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han L, Hipwell JH, Eiben B, Barratt D, Modat M, Ourselin S, Hawkes DJ. A nonlinear biomechanical model based registration method for aligning prone and supine MR breast images. IEEE Trans Med Imaging. 2014 Mar;33(3):682-94. doi: 10.1109/TMI.2013.2294539. PMID 24595342
- [Background] Han L, Hipwell JH, Tanner C, Taylor Z, Mertzanidou T, Cardoso J, Ourselin S, Hawkes DJ. Development of patient-specific biomechanical models for predicting large breast deformation. Phys Med Biol. 2012 Jan 21;57(2):455-72. doi: 10.1088/0031-9155/57/2/455. Epub 2011 Dec 15. PMID 22173131
- [Background] Gefen A, Dilmoney B. Mechanics of the normal woman's breast. Technol Health Care. 2007;15(4):259-71. PMID 17673835
- [Background] Escoffier C, de Rigal J, Rochefort A, Vasselet R, Leveque JL, Agache PG. Age-related mechanical properties of human skin: an in vivo study. J Invest Dermatol. 1989 Sep;93(3):353-7. PMID 2768836
- [Background] Krueger N, Luebberding S, Oltmer M, Streker M, Kerscher M. Age-related changes in skin mechanical properties: a quantitative evaluation of 120 female subjects. Skin Res Technol. 2011 May;17(2):141-8. doi: 10.1111/j.1600-0846.2010.00486.x. Epub 2011 Feb 1. PMID 21281361
- [Background] Kim E, Cho G, Won NG, Cho J. Age-related changes in skin bio-mechanical properties: the neck skin compared with the cheek and forearm skin in Korean females. Skin Res Technol. 2013 Aug;19(3):236-41. doi: 10.1111/srt.12020. Epub 2013 Feb 26. PMID 23441628
- [Background] Ryu HS, Joo YH, Kim SO, Park KC, Youn SW. Influence of age and regional differences on skin elasticity as measured by the Cutometer. Skin Res Technol. 2008 Aug;14(3):354-8. doi: 10.1111/j.1600-0846.2008.00302.x. PMID 19159383
- [Background] Diridollou S, Vabre V, Berson M, Vaillant L, Black D, Lagarde JM, Gregoire JM, Gall Y, Patat F. Skin ageing: changes of physical properties of human skin in vivo. Int J Cosmet Sci. 2001 Dec;23(6):353-62. doi: 10.1046/j.0412-5463.2001.00105.x. PMID 18498486
- [Background] Diridollou S, Black D, Lagarde JM, Gall Y, Berson M, Vabre V, Patat F, Vaillant L. Sex- and site-dependent variations in the thickness and mechanical properties of human skin in vivo. Int J Cosmet Sci. 2000 Dec;22(6):421-35. PMID 18503429
- [Background] Diridollou S, Patat F, Gens F, Vaillant L, Black D, Lagarde JM, Gall Y, Berson M. In vivo model of the mechanical properties of the human skin under suction. Skin Res Technol. 2000 Nov;6(4):214-221. doi: 10.1034/j.1600-0846.2000.006004214.x. PMID 11428960
- [Background] Hendriks FM, Brokken D, van Eemeren JT, Oomens CW, Baaijens FP, Horsten JB. A numerical-experimental method to characterize the non-linear mechanical behaviour of human skin. Skin Res Technol. 2003 Aug;9(3):274-83. doi: 10.1034/j.1600-0846.2003.00019.x. PMID 12877691
- [Background] Kappert KDR, Connesson N, Elahi SA, Boonstra S, Balm AJM, van der Heijden F, Payan Y. In-vivo tongue stiffness measured by aspiration: Resting vs general anesthesia. J Biomech. 2021 Jan 4;114:110147. doi: 10.1016/j.jbiomech.2020.110147. Epub 2020 Nov 25. PMID 33276256
- [Background] Schneider DC, Davidson TM, Nahum AM. In vitro biaxial stress-strain response of human skin. Arch Otolaryngol. 1984 May;110(5):329-33. doi: 10.1001/archotol.1984.00800310053012. PMID 6712522
- [Background] Kvistedal YA, Nielsen PM. Estimating material parameters of human skin in vivo. Biomech Model Mechanobiol. 2009 Feb;8(1):1-8. doi: 10.1007/s10237-007-0112-z. Epub 2007 Nov 27. PMID 18040732
- [Background] Reihsner R, Balogh B, Menzel EJ. Two-dimensional elastic properties of human skin in terms of an incremental model at the in vivo configuration. Med Eng Phys. 1995 Jun;17(4):304-13. doi: 10.1016/1350-4533(95)90856-7. PMID 7633759
- [Background] Sutradhar A, Miller MJ. In vivo measurement of breast skin elasticity and breast skin thickness. Skin Res Technol. 2013 Feb;19(1):e191-9. doi: 10.1111/j.1600-0846.2012.00627.x. Epub 2012 Aug 14. PMID 22891621
- [Background] Coltman CE, Steele JR, McGhee DE. Effect of aging on breast skin thickness and elasticity: implications for breast support. Skin Res Technol. 2017 Aug;23(3):303-311. doi: 10.1111/srt.12335. Epub 2016 Nov 1. PMID 27800637
- [Background] Coumare R, Bouten L, Barbier F. Influence of the menstrual cycle on breast skin elasticity. Comput Methods Biomech Biomed Engin. 2015;18 Suppl 1:1912-3. doi: 10.1080/10255842.2015.1069558. Epub 2015 Aug 14. No abstract available. PMID 26273846
- [Background] Mira A, Carton AK, Muller S, Payan Y. A biomechanical breast model evaluated with respect to MRI data collected in three different positions. Clin Biomech (Bristol). 2018 Dec;60:191-199. doi: 10.1016/j.clinbiomech.2018.10.020. Epub 2018 Oct 17. PMID 30408760
- [Result] Duraes M, Briot N, Connesson N, Chagnon G, Payan Y, Duflos C, Rathat G, Captier G, Subsol G, Herlin C. Evaluation of breast skin and tissue stiffness using a non-invasive aspiration device and impact of clinical predictors. Clin Anat. 2024 Apr;37(3):329-336. doi: 10.1002/ca.24134. Epub 2024 Jan 4. PMID 38174585
- [Derived] Duraes M, Rathat G, Coutureau J, Mandoul C, Francini S, Rebel L, Captier G, Subsol G, Herlin C. New Insights on Breast Anatomy Based on Magnetic Resonance Imaging and Surgical Observations. Clin Anat. 2026 Jan 19. doi: 10.1002/ca.70071. Online ahead of print. PMID 41549904
- See also: Suction Chamber Methods for Measurement of Skin Mechanics : The New Digital Version of the Cutometer. — https://researchportal.vub.be/nl/publications/suction-chamber-methods-for-measurement-of-skin-mechanics-the-new
- See also: In-Vivo Soft Tissues Mechanical Characterization: Volume-Based Aspiration Method Validated on Silicones — https://link.springer.com/article/10.1007/s11340-018-00440-9